CLINICAL TRIAL: NCT00733967
Title: A Human Laboratory Assessment of the Safety and Potential Efficacy of Varenicline In Methamphetamine-Dependent Volunteers Receiving Methamphetamine
Brief Title: Varenicline-Methamphetamine Interaction Study (2008)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No longer active
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Richard De La Garza, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Single Group | Masking: Quadruple
Other Study IDs: H-22707; P50DA018185 (NIH); DPMC (Other: NIDA); 2P50DA018197-06 (NIH)
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Methamphetamine Dependence; Substance Abuse; Methamphetamine Abuse
Keywords: Methamphetamine; Chantix; Varenicline
MeSH Terms: conditions — Substance-Related Disorders | interventions — Varenicline; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Matching oral placebo capsules as control.
  Interventions: Drug: Placebo
- Varenicline (Active Comparator): See assigned interventions.
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — Varenicline (oral capsule): 0.5 mg once daily for 3 days; 0.5 mg twice daily for 2 days; 1 mg twice daily for one day; 1 mg once daily for one day.
  Other Names: Chantix
  Arms: Varenicline
Drug: Placebo — Matching oral placebo capsules as control.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The primary aim of the study is to determine the safety and tolerability of treatment with Varenicline in methamphetamine-dependent volunteers. The investigators also seek to determine the effects of treatment with Varenicline, as compared to placebo, on craving for methamphetamine or cigarettes following exposure to methamphetamine and smoking cues, respectively. The effects of treatment with Varenicline, as compared to placebo, on subjective effects produced by administration of methamphetamine or placebo will be attempted to be determined. Lastly, the investigators hope to determine the effects of treatment with Varenicline, as compared to placebo, on reinforcing effects produced by administration of methamphetamine or placebo.

DETAILED DESCRIPTION:
See Brief Summary

ELIGIBILITY:
Inclusion Criteria:

* English speaking volunteers who are not seeking treatment at the time of the study
* Be between 18-55 years of age
* Meet DSM-IV criteria for MA dependence
* Must be cigarette smokers, defined as smoking 10 or more cigarettes per day by self-report
* Have a self-reported history of using MA by the smoked or IV route and provide at least one MA-positive urine prior to admission
* Have vital signs as follows: resting pulse between 50 and 90 bpm, blood pressures between 105-150 mm Hg systolic and 45-90 mm HG diastolic; this criterion must be met within 2 days of admission
* Have hematology and chemistry laboratory tests that are within normal (+/- 10%) limits with the following exceptions: a) liver function tests (total Bilirubin, ALT, AST, and alkaline phosphatase) < 3 x the upper limit of normal, and b) kidney function tests (creatinine and BUN) < 2 x the upper limit of normal
* Have a baseline EKG that demonstrates normal sinus rhythm, normal conduction (including QTc), and no clinically significant arrhythmias
* Have a medical history and brief physical examination demonstrating no clinically significant contradictions for study participation, in the judgment of the admitting physician or nurse practitioner and the principal investigator

Exclusion Criteria:

* Have any history or evidence suggestive of seizure disorder or brain injury
* Have any previous medically adverse reaction to MA, including loss of consciousness, chest pain, or epileptic seizure
* Have neurological or psychiatric disorders, such as: psychosis, bipolar illness or major depression as assessed by MINI; organic brain disease or dementia assessed by clinical interview; history of any psychiatric disorder which would require ongoing treatment or which would make study compliance difficult; history of suicide attempts within the past three months assessed by MINI and/or current suicidal ideation/plan as assessed by MINI
* Have evidence of clinically significant heart disease or hypertension, as determined by the PI
* Have a family history in first-degree relatives of early cardiovascular morbidity or mortality, as determined by the PI
* Have evidence of untreated or unstable medical illness including: neuroendocrine, autoimmune, renal, hepatic, or active infectious disease
* Have HIV and are currently symptomatic, have a diagnosis of AIDS, or are receiving antiretroviral medication
* Be pregnant or nursing. Other females must either be unable to conceive (i.e., surgically sterilized, sterile, or post-menopausal) or be using a reliable form of contraception (e.g., abstinence, birth control pills, intrauterine device, condoms, or spermicide). All females must provide negative pregnancy urine tests before study entry, upon hospital admission, and at the end of study participation
* Have asthma or currently use alpha or beta agonists, theophylline, or other sympathomimetics
* Have any other illness, condition, or use of psychotropic medications, which in the opinion of the PI and/or the admitting physician or nurse practitioner would preclude safe and/or successful completion of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Effects of varenicline and methamphetamine on cardiovascular measures.
  The safety of MA administration during treatment will be assessed by reporting of adverse events (AEs), and using ECG recording, and heart rate and blood pressure measurements. Digital 12-lead EKG will also be recorded prior to randomization. Blood pressure and heart rate will be measured from 15 min prior to MA or placebo dosing until 2 h after dosing. In addition, heart rate and blood pressure will be assessed throughout the inpatient portion of the protocol.

SECONDARY OUTCOMES:
Effects of varenicline and methamphetamine on subjective measures
  Efficacy will be assessed by measuring effects of treatment on subjective and reinforcing effects produced by administration of MA and craving produced by exposure to drug cues. Other diagnostic measures and assessment instruments will be used to further characterize the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Richard De La Garza, II, PhD, Principal Investigator — Baylor College of Medicine